CLINICAL TRIAL: NCT00948207
Title: Online Narrative Interventions and Family Support for Advanced Cancer Patients
Brief Title: Online and Narrative Interventions for Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M-2009-1189; R21CA129890-01A2 (NIH); CC09310 (Other: University of Wisconsin Carbone Cancer Center); M-2009-1189 (Other: Institutional Review Board); A568000 (Other: UW Madison); PHARM/SRC (Other: UW Madison)
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2016-02

CONDITIONS: Metastatic Cancer
Keywords: Metastatic Cancer; Recurrent Cancer; Distributed Hematological Cancer; Advanced Cancer; Terminal Cancer; Stage III Cancer; Stage IV Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- My Living Story (Experimental): "My Living Story" elicits a dignity-enhancing life story via a telephone interview, and delivers the edited transcript on the patient's personal miLivingStory social network. miLivingStory also provides a direct link to miStory, a life review education website with links to high quality websites that provide cancer information, databases to "do your own research", social support, interactive planning tools, and a page to add their own weblinks.
  miLivingStory and miStory are both password protected.
  Interventions: Behavioral: My Living Story
- My Own Resources (Active Comparator): My Own Resources offers usual care access to high quality websites that provide cancer information, databases to "do your own research," social support, and interactive planning tools. Participants will receive access to the website miOwnResources.
  Interventions: Behavioral: My Living Story; Behavioral: My Own Resources

INTERVENTIONS:
Behavioral: My Living Story — Components include:
  1. Life Review Interview by phone (questions based on Chochinov, 2002 dignity enhancing interview);
  2) Edited transcript is delivered in a word format on...;
  3) miLivingStory, a personal social network, where participants can manage content, design and layer; invite and manage their fiends and family.
  4) miStory, a life review education website and portal to websites for: cancer information, databases to "do your own research," social support, interactive planning tools, and a page to add their own weblinks.
Behavioral: My Own Resources — miOwnResources is a personalized, password-protected web portal to high quality websites that provide cancer information, cancer research databases for "do your own research," social support, and interactive planning tools. miOwnResources also has a page for participants to add their own weblinks.
  Arms: My Own Resources

SUMMARY:
The investigators will test whether narrative life review and web-based social networking for middle aged adults with advanced cancer will improve:

1. existential well being (and reduce psychological distress)
2. generativity and relationship quality, thereby mediating the intervention effects

The investigators will also conduct exploratory process analyses of each participant's social network.

DETAILED DESCRIPTION:
Middle aged patients with advanced cancer report more distress, and active search for meaning and personal growth than older and/or early stage patients. Nonetheless, such positive growth is far from typical and interventions help. Expert-guided life review reduced distress for hospice patients, but is not widely accessible-and many patients lack the energy or skill to write their own life story. Online cancer information and support expert systems improve quality of life. Patients are increasingly developing their own social networks, but many lack the skills to do so. Moreover the effects on social networking on patient well-being have not been studied.

"My Living Story" elicits a dignity-enhancing life story via a telephone interview (based on Chochinov, JAMA 2002), and delivers the edited transcript on the patient's personal miLivingStory social network. miLivingStory links to a life review education website (called miStory) with links to high quality cancer information, support and interactive planning tools.

We hypothesize that telling, revising and sharing the life story with one's selected social network will improve the patient's existential well-being and reduce their distress. Furthermore, we hypothesize that these effects will be mediated by My Living Story's effects on improving the patient's sense of legacy (generativity) and the quality of their relationships. Our exploratory observational analyses of each individual miLivingStory network will contribute to an understanding of how social network configuration and communication patterns correlate with measured outcomes

We will recruit and randomize 100 patients with advanced cancer. The control group will receive a personalized web portal (called miOwnResources) with links to high quality cancer information, social support and interactive planning tools, and a feature to add their own links. All participants will sign informed consent forms, complete a pre-test survey and post-tests at tow and four months.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 60,
* Stage III or IV Cancer,
* Able and willing to use an internet computer to complete study activities.

Exclusion Criteria:

* Institutionalized, < 6 months prognosis,
* Cannot read or understand English,
* Unable or unwilling to use an internet computer to complete study activities.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Existential Well-being (FACIT-Sp) | 0, 2 and 4 months

SECONDARY OUTCOMES:
Distress (POMS-SF) | 0, 2, and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret (Meg) E Wise, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu